CLINICAL TRIAL: NCT07173699
Title: Evaluation of the Effect of Salivary Melatonin Levels on Postoperative Pain and Sleep Quality Following Endodontic Treatments Performed at Different Times of Day
Brief Title: Evaluation of the Effect of Salivary Melatonin Levels on Postoperative Pain and Sleep Quality Following Endodontic Treatments Performed at Different Days and Times
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, KEZBAN MELTEM ÇOLAK, KEZBAN MELTEM COLAK, Ataturk University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ATU-ENDO-MELATONIN-2025
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Pain After Endodontic Treatment
Keywords: Root Canal Treatment; Salivary Melatonin; Circadian Rhythm; Postoperative Pain; Sleep Quality
MeSH Terms: conditions — Pain, Postoperative; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Split-mouth crossover design: Each participant will receive root canal treatment on two asymptomatic mandibular molars, one in the morning session and the other in the afternoon session, with a one-week interval.
Masking Description: This is an open-label study; both participants and investigators are aware of the timing of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Morning Arm (Experimental): Root canal treatment performed on an asymptomatic mandibular molar in the morning session (08:30-09:30). Standard endodontic protocol will be applied. Saliva samples will be collected before the procedure for melatonin analysis, and postoperative pain and sleep quality will be assessed.
  Interventions: Procedure: root canal treatment
- Arm 2: Afternoon Arm (Experimental): Root canal treatment performed on an asymptomatic mandibular molar in the afternoon session (14:00-15:00). Standard endodontic protocol will be applied. Saliva samples will be collected before the procedure for melatonin analysis, and postoperative pain and sleep quality will be assessed.
  Interventions: Procedure: root canal treatment

INTERVENTIONS:
Procedure: root canal treatment — Standardized root canal treatment performed on asymptomatic mandibular molars. Procedures include local anesthesia, rubber dam isolation, access cavity preparation, cleaning and shaping with rotary instruments, irrigation with NaOCl and EDTA, and obturation using a standardized protocol. Saliva samples are collected prior to treatment for melatonin analysis. Postoperative pain and sleep quality are assessed using validated questionnaires.

SUMMARY:
This clinical study aims to evaluate the effect of salivary melatonin levels on postoperative pain and sleep quality in patients undergoing root canal treatment at different times of the day. Each participant will receive endodontic treatment on two asymptomatic mandibular molars, one in the morning and the other in the afternoon. Pain intensity and sleep quality will be assessed using standard questionnaires, and salivary melatonin levels will be analyzed.

DETAILED DESCRIPTION:
Postoperative pain following endodontic treatment is a common clinical problem that adversely affects patients' quality of life. Studies have shown that this pain may not only be associated with local tissue trauma and inflammation but can also vary depending on the individual's neuroendocrine system and biological clock (Alhassani & AlGhamdi, 2021).

Many physiological processes in the human body are regulated by the circadian rhythm, which directly influences pain perception, inflammatory responses, and hormone secretion (Smolensky et al., 2015). One of the primary regulatory hormones of circadian rhythm is melatonin, which is secreted mainly by the pineal gland as well as other tissues, reaching peak levels particularly during nighttime. Melatonin is known for its analgesic, anti-inflammatory, antiproliferative, and immunomodulatory properties (Reiter et al., 2010).

In recent years, the effects of melatonin in dentistry have been investigated in the contexts of periodontal regeneration, oral mucosal healing, and bone regeneration (Cutando et al., 2007; Dominguez-Rodriguez et al., 2010). However, clinical studies exploring the role of melatonin during endodontic treatment and its influence on postoperative pain remain very limited. Similarly, no studies in the literature have specifically examined the relationship between melatonin levels and sleep quality in the context of endodontic therapy.

Moreover, some research suggests that dental procedures performed at different times of the day may have varying effects on postoperative pain intensity and the healing process (Segura-Egea et al., 2008). In this regard, understanding how endodontic treatment interacts with systemic biological processes when performed at different times of day is clinically significant.

This study will analyze salivary melatonin levels obtained prior to morning and afternoon endodontic procedures performed on the same patient and will subsequently evaluate their relationship with postoperative pain levels and sleep quality. In doing so, it will provide some of the first clinical evidence regarding the impact of circadian rhythm and melatonin on pain and sleep following endodontic treatment.

In this way, the study not only offers an original approach that may guide clinical practice but also has the potential to lay the groundwork for a personalized dental treatment concept aligned with biological rhythms.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 25-45 years Patients with two asymptomatic, devital mandibular molars in the same arch No radiographic evidence of periapical lesions or pathological formations in the teeth Patients without systemic diseases (ASA I) Patients who have not used antibiotics, analgesics, or melatonin-containing medications within the last week Patients who have signed the informed consent form

Exclusion Criteria:

Patients with a diagnosis of sleep disorder or those regularly using sleep medications/sedatives Patients with systemic diseases (e.g., hypertension, diabetes, endocrine disorders, etc.) Patients receiving psychiatric treatment Pregnant or breastfeeding patients Patients unable to cooperate during the treatment process Patients with restorative or periodontal complications in their teeth Patients working in a shift system

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity | Within 7 days after each root canal treatment session
  Pain intensity will be assessed using a 10-cm Visual Analogue Scale (VAS), where 0 represents "no pain" and 10 represents "worst pain imaginable." Participants will record their pain levels following root canal treatment sessions performed in the morning and afternoon.

SECONDARY OUTCOMES:
Sleep quality | Within 7 days after each root canal treatment session
  Sleep quality will be evaluated using the Pittsburgh Sleep Quality Index (PSQI). The PSQI measures subjective sleep quality over the past month, but in this study, patients will complete it for the week following each root canal treatment session (morning and afternoon).

CONTACTS AND LOCATIONS:
Overall Officials: KEZBAN MELTEM COLAK, PROF., Principal Investigator — Atatürk University, Faculty of Dentistry, Department of Endodontics
Locations (1):
- Atatürk University Faculty of Dentistry, Department of Endodontics, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a single-center academic thesis study with a limited number of patients. Data include personal health information, and sharing outside the study team is restricted due to ethical and confidentiality considerations.

REFERENCES:
- [Background] Benloucif S, Burgess HJ, Klerman EB, Lewy AJ, Middleton B, Murphy PJ, Parry BL, Revell VL. Measuring melatonin in humans. J Clin Sleep Med. 2008 Feb 15;4(1):66-9. PMID 18350967
- [Background] Segura-Egea JJ, Cisneros-Cabello R, Llamas-Carreras JM, Velasco-Ortega E. Pain associated with root canal treatment. Int Endod J. 2009 Jul;42(7):614-20. doi: 10.1111/j.1365-2591.2009.01562.x. Epub 2009 May 8. PMID 19467050